CLINICAL TRIAL: NCT02010632
Title: Comparative Pharmacodynamics and Pharmacokinetics Study of Generic and Reference Clopidogrel Products in Thai Healthy Volunteers
Brief Title: Comparative Pharmacodynamics and Pharmacokinetics Study of Generic and Reference Clopidogrel Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Wichittra Tassaneeyakul, Professor Dr. Wichittra Tassaneeyakul, Departments of Pharmacology, Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: PDPK-CLO-2013
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Pharmacodynamics
Keywords: Clopidogrel; Platelet inhibition; Platelet aggregation
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Generic clopidogrel product (Experimental): Apolets® 75 mg tablet
  Interventions: Drug: Generic clopidogrel product Apolets®
- Original clopidogrel product (Active Comparator): Plavix® 75mg tablet
  Interventions: Drug: Original clopidogrel product Plavix®

INTERVENTIONS:
Drug: Generic clopidogrel product Apolets® — * Clopidogrel 75 mg once daily for 7 days
  * Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
  Other Names: Apolets®
  Arms: Generic clopidogrel product
Drug: Original clopidogrel product Plavix® — * Clopidogrel 75 mg once daily for 7 days
  * Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
  Other Names: Plavix®
  Arms: Original clopidogrel product

SUMMARY:
The purpose of this study is to compare the pharmacodynamic effect of clopidogrel on the platelet inhibition and the pharmacokinetic profiles of clopidogrel carboxylic acid metabolite between generic and reference clopidogrel products in Thai healthy volunteers

DETAILED DESCRIPTION:
Platelet aggregation (ex vivo) were measured by using Whole blood impedence aggregometry (Chrono-log®) and VerifyNow® P2Y12 assay. Plasma concentration of clopidogrel carboxylic acid metabolite were measured by High performance liquid chromatography (HPLC).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Body mass index between 18-25 kg/m2
* No clinically significant abnormalities, as confirmed on medical history; detailed physical examination; clinical laboratory analysis (blood hematology, biochemistry, prothrombin time, bleeding time, and urinalysis)

Exclusion Criteria:

* An allergy to any drug; and/or a history of drug and/or alcohol abuse.
* Subjects who had donated blood within 3 months prior to the start of this study or had participated in another investigational drug study within 3 months prior to the start of this study
* Participating subjects were instructed to abstain from the use of any drugs for at least 2 weeks before and throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wichittra Tassaneeyakul, Ph.D., Principal Investigator — Khon Kaen University; Somsak Tiamkao, MD, Principal Investigator — Khon Kaen University; Sirimas Kanjanawart, Ph.D., Principal Investigator — Khon Kaen University; Kutcharin Phunikhom, MD, Principal Investigator — Khon Kaen University; Nontaya Nakkam, B.Pharm, Principal Investigator — Khon Kaen University; Thanawat Kaewkamsorn, M.Sc., Principal Investigator — Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khonkaen, Changwat Khon Kaen, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Generic Clopidogrel Product: Apolets® 75 mg tablet (Generic Clopidogrel Product first, wash out period for 14 days then Original Clopidogrel Product) Generic clopidogrel product Apolets®: -Clopidogrel 75 mg once daily for 7 days
  -Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
- Original Clopidogrel Product: Plavix® 75mg tablet (Original Clopidogrel Product first, wash out period for 14 days then Generic Clopidogrel Product) Original clopidogrel product Plavix®: -Clopidogrel 75 mg once daily for 7 days
  -Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
Period: First Intervention (7 Days)
Arm/Group | Generic Clopidogrel Product | Original Clopidogrel Product
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Wash Out Period (14 Days)
Arm/Group | Generic Clopidogrel Product | Original Clopidogrel Product
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Generic Clopidogrel Product | Original Clopidogrel Product
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: First intervention: Apolets® 75 mg tablet (Generic Clopidogrel Product first, wash out period for 14 days then Original Clopidogrel Product) Generic clopidogrel product Apolets®: -Clopidogrel 75 mg once daily for 7 days. Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7 Wash out period: 14 days Second intervention: Plavix® 75mg tablet (Original Clopidogrel Product first, wash out period for 14 days then Generic Clopidogrel Product) Original clopidogrel product Plavix®: -Clopidogrel 75 mg once daily for 7 days. Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.43 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Region of Enrollment [Number; unit: participants]
  Thailand | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.12 (2.75)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamic Effect: The Platelet Inhibition Effect of Clopidogrel at the Various Times on Day 7 (0-24 Hours) (at Steady State)
Time Frame: Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
Measure: Mean (Standard Deviation); unit: percent inhibition*hour
Groups:
- Generic Clopidogrel Product: Apolets® 75 mg tablet
  Generic clopidogrel product Apolets®: -Clopidogrel 75 mg once daily for 7 days
  -Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
- Original Clopidogrel Product: Plavix® 75mg tablet
  Original clopidogrel product Plavix®: -Clopidogrel 75 mg once daily for 7 days
  -Blood collection at 0 (before dosing), 1, 2, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
Arm/Group | Generic Clopidogrel Product | Original Clopidogrel Product
Number analyzed (Participants) | 31 | 31
percent inhibition*hour | 1853.58 (673.95) | 1892.84 (657.22)

2. Secondary Outcome: Pharmacokinetic Profiles: Area Under the Concentration-Time Curve (AUC 0-24)
Time Frame: Blood collection at 0 (before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours after the last dose, administered at day 7
Reporting Status: Not Posted

3. Secondary Outcome: Pharmacokinetic Profiles: The Maximum Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetic Profiles: Time to Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Generic Clopidogrel Product | Original Clopidogrel Product
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No